CLINICAL TRIAL: NCT06752681
Title: A Phase 1, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of the PTK7-Targeted Antibody-drug Conjugate DAY301 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of DAY301 in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Day One Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAY301-001
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: Advanced or metastatic solid tumors; Dose Escalation; Dose Expansion; DAY301; PTK7-Targeted Antibody-drug Conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DAY301 intravenous (IV) infusion (Experimental): DAY301 will be administered at different dose levels in dose escalation and at the RD in dose expansion cohorts.
  Interventions: Drug: DAY301

INTERVENTIONS:
Drug: DAY301 — DAY301 will be administered as IV infusion

SUMMARY:
This is a Phase 1a/1b, open-label, dose escalation and expansion study to evaluate the safety and anti-tumor activity of DAY301, a PTK7-directed antibody-drug conjugate in participants with advanced or metastatic solid tumors. The study comprises of 2 phases: Phase 1a dose escalation where participants will be administered DAY301 at escalating dose levels to assess safety and tolerability, and to determine the maximum tolerated dose (MTD) and/or the recommended dose (RD); In Phase 1b dose expansion, DAY301 will be evaluated in dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors of the following histologies:
* Ovarian cancer
* Esophageal squamous cell carcinoma
* Triple-negative breast cancer
* Non-small cell lung cancer
* Small cell lung cancer
* Head and neck squamous cell carcinoma
* Gastric/gastroesophageal junction adenocarcinoma
* Cervical squamous cell carcinoma
* Endometrial cancers

(Participants must have been previously treated with standard of care systemic therapy, or for whom no standard therapy is available).

* Availability of tumor tissue sample (either an archival specimen or a fresh biopsy) at screening
* Measurable disease per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Prior use of PTK7 targeting treatment (Phase 1a) or prior use of PTK7 targeting treatments and/or topoisomerase 1 (TOP1) inhibitor-based antibody-drug conjugate (ADC) (Phase 1b).
* Phase 1b disease-specific exclusion criteria:

  1. Cohort 1: Neuroendocrine tumors or endometrial sarcoma (eg, stromal sarcoma, leiomyosarcoma, or other types of pure sarcomas)
  2. Cohort 2: Ovarian cancer that progressed >6 months after the last dose of platinum-based chemotherapy (platinum-sensitive disease), or disease that did not respond (partial response [PR] or complete response [CR]) to or progressed ≤91 days after the last dose of first-line platinum-based chemotherapy (primary platinum-refractory disease)
  3. Cohort 3: nasopharyngeal primary tumors.
* History of small bowel obstruction requiring hospitalization within 3 months prior to the first dose of study treatment.
* Ascites requiring frequent paracentesis (more often than approximately every 4 weeks) for symptomatic management, or new onset within 4 weeks prior to the first dose of study treatment. Patients with an indwelling catheter may be considered eligible, after consultation with the medical monitor.
* Active or progressing brain metastases or evidence of leptomeningeal disease.
* Persistent toxicities from previous systemic antineoplastic treatments of Grade >1, excluding alopecia and vitiligo.
* Systemic antineoplastic therapy within five half-lives or 4 weeks, whichever is shorter, prior to first dose of study treatment, including investigational agents.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Dose Escalation: Number of participants with reported Dose Limiting Toxicities (DLTs) | Within 21 days of first infusion (Day 1)
  To evaluate adverse events (AEs) considered dose limiting toxicities that occur in the first cycle of treatment (within a DLT observation period).
Phase 1a: Dose Escalation: Number of participants with reported adverse events (AEs) or serious AEs (SAEs) | through the duration of treatment, up to approximately 12 months
  The type, incidence, and severity of AEs and SAEs will be determined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Phase 1a: Dose Escalation: Frequency of dose interruptions | through the duration of treatment, up to approximately 12 months
  The frequency at which dose interruptions occur during dose-escalation
Phase 1a: Dose Escalation: Duration of dose interruptions | through the duration of treatment, up to approximately 12 months
  The duration of dose interruptions that occur during dose-escalation.
Phase 1a: Dose Escalation: Frequency of dose reductions | through the duration of treatment, up to approximately 12 months
  The frequency at which dose reductions occur during dose-escalation.
Phase 1a: Dose Escalation: Duration of dose reductions | through the duration of treatment, up to approximately 12 months
  The duration of dose reductions that occur during dose-escalation.
Phase 1b: Dose Expansion: Objective response rate | through the duration of treatment, up to approximately 12 months-up
  Objective response rate based on best overall response (BOR) will be assessed by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Phase 1b: Dose Expansion: Number of participants reporting AEs and SAEs | through the duration of treatment, up to approximately 12 months
  The type, incidence, and severity of AEs and SAEs will be determined using the NCI CTCAE v5.0.
Phase 1b: Dose Expansion: Frequency of dose interruptions | through the duration of treatment, up to approximately 12 months
  The frequency at which dose interruptions occur during dose-expansion.
Phase 1b: Dose Expansion: Duration of dose interruption | through the duration of treatment, up to approximately 12 months
  The duration of dose interruptions that occur during dose-expansion.
Phase 1b: Dose Expansion: Frequency of dose reductions | through the duration of treatment, up to approximately 12 months
  The frequency at which dose reductions occur during dose-expansion.
Phase 1b: Dose Expansion: Duration of dose reductions | through the duration of treatment, up to approximately 12 months
  The duration of dose reductions that occur during dose-expansion.

SECONDARY OUTCOMES:
Phase 1a and Phase 1b: Maximum concentration (Cmax) of DAY301 | Varying timepoints through the duration of treatment, up to approximately 12 months
  Blood samples will be collected at indicated time points for the analysis of pharmacokinetic parameters.
Phase 1a and Phase 1b: time to Cmax (Tmax) of DAY301 | Varying timepoints through the duration of treatment, up to approximately 12 months
  Blood samples will be collected at indicated time points for the analysis of pharmacokinetic parameters.
Phase 1a and Phase 1b: area under the curve (AUC) of DAY301 | Varying timepoints through the duration of treatment, up to approximately 12 months
  Blood samples will be collected at indicated time points for the analysis of pharmacokinetic parameters.
Phase 1a and Phase 1b: terminal half-life (t1/2) of DAY301 | Varying timepoints through the duration of treatment, up to approximately 12 months
  Blood samples will be collected at indicated time points for the analysis of pharmacokinetic parameters.
Phase 1a Dose Escalation: Objective response rate | through the duration of treatment, up to approximately 12 months
  Objective response rate based on BOR will be assessed by investigators according to RECIST v1.1.
Phase 1a and 1b: Clinical Benefit rate (CBR) | through the duration of treatment, up to approximately 12 months
  Clinical Benefit rate will be assessed by investigators according to RECIST v1.1.
Phase 1a and 1b: duration of response (DOR) | through the duration of treatment, up to approximately 12 months
  Duration of response will be assessed by investigators according to RECIST v1.1.
Phase 1a and 1b: time to response (TTR) | through the duration of treatment, up to approximately 12 months
  Time to response will be assessed by investigators according to RECIST v1.1.
Phase 1a and 1b: Progression-free survival | through the duration of treatment, up to approximately 12 months
  Progression-free survival will be assessed by investigators according to RECIST v1.1.
Phase 1b: Overall survival | through the duration of treatment, up to approximately 12 months
  Overall survival will be assessed by investigators.
Phase 1a and 1b: Number of participants with positive antidrug antibodies (ADAs) | varying timepoints through the duration of treatment, up to approximately 12 months
  Assessed by the measure of anti-drug antibodies in serum.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Site: 001-058, New Haven, Connecticut
  - Site: 001-063, Lake Mary, Florida
  - Site: 001-064, Sarasota, Florida
  - Site: 001-060, Indianapolis, Indiana
  - Site: 001-059, Grand Rapids, Michigan
  - Site: 001-039, New York, New York
  - Site: 001-073, Oklahoma City, Oklahoma
  - Site: 001-065, Nashville, Tennessee
  - Site: 001-069, Houston, Texas
  - Site: 001-057, San Antonio, Texas
- Canada (2):
  - Site: 011-013, Vancouver, British Columbia
  - Site: 011-005, Toronto, Ontario